CLINICAL TRIAL: NCT02074943
Title: Efficacy and Safety of Platelet Rich Plasma in Androgenetic Alopecia: A Double-Blind, Randomized, Placebo Controlled Trial
Brief Title: Efficacy and Safety of Platelet Rich Plasma in Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Jerry Shapiro, Clinical Professor, Vancouver General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H13-03126
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRP/Saline (Experimental): Same patient will be injected with PRP and normal saline. Each one will be inject on half head.
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — PRP will be inject to half head. The other half will be injected with normal saline.

SUMMARY:
The investigators plan to conduct a clinical trial to assess the effects and safety of platelet rich plasma on androgenetic alopecia.

DETAILED DESCRIPTION:
Platelet rich plasma (PRP) is made from your own blood by taking a sample of venous blood, placing it in a special tube, and spinning the blood in a centrifuge which is a piece of equipment used to separate the components of blood. Blood is made of red blood cells, white blood cells and platelets, while plasma, the liquid component is predominantly water but also contains clotting factors, proteins, and glucose. Platelets are small, disk shaped clear cell fragments which are a natural source of growth factors. They circulate in the blood and are involved in hemostasis which is a process which causes bleeding to stop, leading to the formation of blood clots. So-called "Platelet-rich plasma" represents the patient's own plasma that has been mechanically centrifuged to increase the concentration of platelets compared to the whole blood. The basic idea behind PRP injection is to deliver high concentrations of growth factors to the scalp, with the hope of stimulating hair regrowth.

PRP is an innovative therapy and has been used since 1987 to help promote healing in orthopedic surgery, dental surgery and dermatology. Recently, there have been reports supporting the use of PRP in the treatment of hair loss.

Androgenetic alopecia (AGA) is the most common cause of hair loss. It has very limited treatment modalities which includes minoxidil, 5-alpha reductase inhibitors and hair transplantation. Each option has its own side effects range from hypertrichosis which is excessive hair growth, possible birth defects if given to women of child bearing age, decreased libido and the possibility of prolonged impotence.

To our best knowledge, there are no double blind, randomized, placebo-controlled trials evaluating the efficacy and safety of PRP injection in treating AGA. A placebo is a simulated or otherwise medically ineffectual treatment for a disease or other medical condition intended to deceive the recipient. The investigators plan to conduct a clinical trial to assess the effects and safety of PRP on AGA. The investigators also plan to identify the presence of various growth factors in PRP and their correlations in hair regrowth.

ELIGIBILITY:
Inclusion Criteria:

* Males and females in good general health, ages 18-70.
* Patients with mild to moderate AGA (Ludwig alopecia score I and II, and the Hamilton-Norwood score 1 to 4).

Exclusion Criteria:

* Patients who received treatments for AGA within the last 3 months.
* Patients who have active or history of malignancies.
* Patients with platelets disorders, anemia and or bleeding disorders.
* Women who are pregnant or breast-feeding.
* Un-cooperative patients or patients who are unable to understand the protocol or give informed consent.
* Patients who are known to be HIV, hepatitis B or C positive or otherwise immunocompromised.
* Subjects who have active skin disease or skin infection at the intended treatment area.
* Patients on non-steroidal anti-inflammatory medications.
* Patients with a propensity for keloids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The degree of hair regrowth based on the hair regrowth score (RGS) for each side of scalp. | 16 weeks

SECONDARY OUTCOMES:
Changes in hair count and caliber. Changes in hair count and caliber | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MD, Principal Investigator — Professor
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, Canada

REFERENCES:
- [Derived] Siah TW, Guo H, Chu T, Santos L, Nakamura H, Leung G, Shapiro J, McElwee KJ. Growth factor concentrations in platelet-rich plasma for androgenetic alopecia: An intra-subject, randomized, blinded, placebo-controlled, pilot study. Exp Dermatol. 2020 Mar;29(3):334-340. doi: 10.1111/exd.14074. Epub 2020 Feb 7. PMID 31984508